CLINICAL TRIAL: NCT02777944
Title: Motivate: A Web Based Intervention to Increase Attendance at an Eating Disorder Service
Brief Title: Motivate: A Web-based Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Collaborators: Dorset HealthCare University NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PhDDay
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Results first posted 2019-07-31 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Eating Disorders
Keywords: motivation; attendance
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Access to Motivate: a web-based intervention, in addition to Usual Care
  Interventions: Behavioral: Motivate: a web-based intervention
- Control (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Motivate: a web-based intervention — A web-based intervention focuses on managing expectations of assessment, addressing ambivalence and increasing users' motivation and confidence to attend their initial appointment. This is achieved through the use of information, motivational tools, interactive activities and stories from other individuals with EDs spread across four 15-20 minute modules.
  Arms: Intervention

SUMMARY:
The aim of this study is to test whether MotivATE can increase attendance at assessment. This will be done using a single-consent Zelen randomised control trial, with all non-emergency adult clients referred to the Kimmeridge Courte Eating Disorder Service over a one year period being randomised to either treatment as usual (TAU) or TAU plus access to the MotivATE intervention prior to their assessment appointment.

DETAILED DESCRIPTION:
MotivATE is a web-based intervention intended to be delivered at the point of referral to an Eating Disorder (ED) service. The intervention focuses on managing expectations of assessment, addressing ambivalence and increasing users' motivation and confidence to attend their initial appointment. This is achieved through the use of information, motivational tools, interactive activities and stories from other individuals with EDs spread across four 15-20 minute modules. These modules have been evaluated by service-users who have an ED.

The aim of this study is to test whether MotivATE can increase attendance at assessment. This will be done using a single-consent Zelen randomised control trial, with all non-emergency adult clients referred to the Kimmeridge Courte Eating Disorder Service over a one year period being randomised to either treatment as usual (TAU) or TAU plus access to the MotivATE intervention prior to their assessment appointment.

Routine audit data will be collected to compare the number of people who attend their assessment appointment in the MotivATE group verses the control group. Usage data generated by the intervention will also be assessed. Twenty participants from the MotivATE group will be invited to give qualitative feedback about their experience of the intervention.

ELIGIBILITY:
Inclusion criteria

1) Referrals to the eating disorders service during the study period.

Exclusion criteria

1. Inpatients or emergency and urgent cases.
2. Patients who have already been randomised into the study.
3. Non English speakers

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Appleton, PhD, Study Director — Bournemouth University

IPD SHARING:
Plan to Share IPD: No
Group data will be publicly available on completion

REFERENCES:
- [Derived] Denison-Day J, Muir S, Newell C, Appleton KM. A Web-Based Intervention (MotivATE) to Increase Attendance at an Eating Disorder Service Assessment Appointment: Zelen Randomized Controlled Trial. J Med Internet Res. 2019 Feb 27;21(2):e11874. doi: 10.2196/11874. PMID 30810533

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 157 | 156
Completed | 157 | 156
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data were not collected, with the exception of geographical region.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 157 | 156 | 313
Age, Customized [Count of Participants; unit: Participants] — Population: Baseline data were not collected.
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Baseline data were not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Participants recruited via referrals to the clinic by General Practitioners
  Participants
    United Kingdom | 157 | 156 | 313

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Attended Initial Assessment Appointment
Description: Attendance at initial assessment appointment
Time Frame: 3 months
Population: Number of participants who attended initial assessment appointment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 157 | 156
Participants | 140 | 134

2. Secondary Outcome: Number of Participants Who Accessed the Intervention Program
Description: Number of participants who accessed the intervention program
Time Frame: 3 months
Population: Number of participants who accessed the intervention program
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 157 | 0
Participants | 53 | 0

3. Secondary Outcome: Number of Participants Who Volunteered to Provide Qualitative Feedback on the Motivate Program
Description: Number of participants who volunteered to provide qualitative feedback on the Motivate Program
Time Frame: 3 months
Population: Qualitative feedback on the intervention program
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 0
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: No data collected
Description: No data collected
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Use of only one site limits the applicability of the findings to general practice.

Lack of a pre-post measure of motivation to change. Potential lack of power in the analysis of the primary research question.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT02777944/Prot_SAP_000.pdf